CLINICAL TRIAL: NCT02417610
Title: Comparative Assessment of Viscosupplementation With Polynucleotides and Hyaluronic Acid to Viscosupplementation With Hyaluronic Acid in the Treatment of Osteoarthritis of the Knee. Randomized, Double-blind, Controlled Study
Brief Title: Comparative Assessment of Viscosupplementation With Polynucleotides and Hyaluronic Acid
Acronym: PNHA1401
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Carubbi, MD, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22/14
Record Dates: First submitted 2015-02-17; First posted 2015-04-15 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis
Keywords: Polynucleotide; Hyaluronic acid; Intra articular injection
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polynucleotide - PNHA - Newart (Experimental): 50 patients will be enrolled and treated with three weekly injections of polynucleotide plus hyaluronic acid
  Interventions: Device: Polynucleotide - PNHA - Newart
- Hyaluronic acid - HA - Ialart (Active Comparator): 50 patients will be enrolled and treated with three weekly injections of hyaluronic acid
  Interventions: Device: Hyaluronic acid - HA - Ialart

INTERVENTIONS:
Device: Polynucleotide - PNHA - Newart — gel polynucleotides and hyaluronic acid
  Arms: Polynucleotide - PNHA - Newart
Device: Hyaluronic acid - HA - Ialart — Hyaluronic acid
  Arms: Hyaluronic acid - HA - Ialart

SUMMARY:
The purpose of the study is to assess the validity of the polynucleotide within the intra articular treatment of osteoarthritis of the knee, comparing it with that of hyaluronic acid, the most commonly used.

DETAILED DESCRIPTION:
This study is double-blind, controlled, randomized.The aim of the study is to evaluate the efficacy, safety and tolerability of polynucleotides and hyaluronic acid gel (PNHA, class III medical device) for intra-articular infiltration in treating pain in osteoarthritis (OA) patients knee.

This study will involve patients with osteoarthritis who comply with the inclusion and exclusion criteria. One hundred patients between the ages of 45 and 70 will be enrolled in the study and randomized to receive one of the following treatment groups:

Group A) Polynucleotides and Hyaluronic Acid (PNHA) Group B) Hyaluronic Acid (HA) The treatment will be administered through intra-articular infiltration, a weekly infiltration in the affected knee, for a total of 3 infiltrations (T0, T1 and T2).

The use of non-steroidal anti-inflammatory drugs (NSAIDs) was permitted, but the use of paracetamol 1 cp 1000 mg every 12 hours, or Meloxicam 15 mg a tablet after meals every 12 hours, was recommended.

In case of grug taking: the number of days when the patient used NSAIDs, the commercial name and the NSAID dosage used were reported in the CRF.

Study visit:

* T0 start study: inclusion in the clinical trial and assignment of the randomization number; radiography; clinical study start-up evaluation; fill in the WOMAC questionnaire; infiltration No. 1.
* T 1 after 1 week from the beginning of the study: infiltration No. 2.
* T 2 after 2 weeks from the beginning of the study (end of treatment): infiltration No. 3.

FOLLOW UP:

* T 3 after 2 months from the beginning of the study: clinical evaluation; fill in the WOMAC questionnaire.
* T 4 after 6 months from the start of the study: clinical evaluation; fill in the WOMAC questionnaire.
* T 5 after 1 year from the beginning of the study: clinical evaluation; fill in the WOMAC questionnaire.
* T 6 after 2 years from the beginning of the study: radiography; clinical evaluation; fill in the WOMAC questionnaire.

At T6 visit, the patient completed the study. A 24-month study period is calculated for each patient.

Any adverse event that occurred during the study period was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 75 years
* Patients informed consent
* Knee OA (Osteoarthritis) (ACR classification) with a Kellgren Laurence from 1 to 4
* Knee pain from arisen at least 2 months
* BMI lower than 40

Exclusion Criteria:

* Pregnancy or lactation
* Severe systemic disorders
* History of drug abuse or alcoholism
* Hypersensibility to Hyaluronic acid or Polynucleotide
* No previous intra articular infiltration (from 3 months)
* No steroidal or anticoagulant systemic therapy from one month
* Knee articular deformity
* Patients affected by rheumatoid arthritis or other inflammatory articular pathologies and hematological disorders
* Focal skin lesion in the anatomical site of injections

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) | 6 months
  The WOMAC is a self-administered questionnaire consisting of 24 items divided into 3 subscales Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
KSS (Knee society score) | 6 months
  The Knee Society Score it comprises two parts, the first addressing pain, stability and range of movement. The second part examines function, with particular reference to walking distance and stair climbing. Maximum scores of 100 are possible in each section, consider a negitive outcome as zero.
  Grading for the knee Society Score
  Excellent: Score 80-100 Good: Score 70-79 Fair: Score 60-69 Poor: Score below 60. A Knee Society Score questionnaire will be used in the study.
Synovial fluid analysis | 3 weeks
  Morphological analysis and blood white cell count
Growth factor contained in synovial fluid determinations | 3 weeks
  Total protein content, IL1beta, IL6, IL8, TNFalpha, MMP1

CONTACTS AND LOCATIONS:
Overall Officials: Dante Dallari, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Derived] Stagni C, Rocchi M, Mazzotta A, Del Piccolo N, Rani N, Govoni M, Vivarelli L, Veronesi F, Fini M, Dallari D. Randomised, double-blind comparison of a fixed co-formulation of intra-articular polynucleotides and hyaluronic acid versus hyaluronic acid alone in the treatment of knee osteoarthritis: two-year follow-up. BMC Musculoskelet Disord. 2021 Sep 12;22(1):773. doi: 10.1186/s12891-021-04648-0. PMID 34511091